CLINICAL TRIAL: NCT06784843
Title: Dexmedetomidine Versus Midazolam as an Adjuvant to Local Anesthetic Mixture (Bupivacaine, Lidocaine, and Hyaluronidase) for Peribulbar Block During Cataract Surgery: A Randomized Controlled Trial
Brief Title: Dexmedetomidine Versus Midazolam for Peribulbar Block
Acronym: peribulbar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, assistant professor, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: peribulbar block
Record Dates: First submitted 2024-12-28; First posted 2025-01-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Cataract
Keywords: dexmedetomidine; midazolam; peribulbar block; cataract
MeSH Terms: conditions — Cataract | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Intervention Model Description: 2 groups
Who Masked: Participant, Care Provider
Masking Description: The allocation sequence was concealed using sealed opaque envelopes . Patients and the operators were masked to the allocation of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- peribulbar block 1 (Active Comparator): Patients who were scheduled for cataract surgery under peribulbar block.
  Interventions: Drug: Dexmedetomidine as an adjuvant to local anesthesia for peribulbar block
- peribulbar block 2 (Active Comparator): Patients who were scheduled for cataract surgery under peribulbar block.
  Interventions: Drug: Midazolam as an adjuvant to local anesthesia for peribulbar block

INTERVENTIONS:
Drug: Dexmedetomidine as an adjuvant to local anesthesia for peribulbar block — Dexmedetomidine as an adjuvant to a local anesthetic mixture (bupivacaine, lidocaine, and hyaluronidase) for peribulbar block during cataract surgery
  Other Names: DEX
  Arms: peribulbar block 1
Drug: Midazolam as an adjuvant to local anesthesia for peribulbar block — Midazolam as an adjuvant to a local anesthetic mixture (bupivacaine, lidocaine, and hyaluronidase) for peribulbar block during cataract surgery
  Other Names: MID
  Arms: peribulbar block 2

SUMMARY:
50 patients of both sexes, ages 18 to 75, who were scheduled for cataract surgery and had physical status I or II according to the American Society of Anesthesiologists were included in this study.

After induction of general anesthesia, all patients received peribulbar block. In group A (midazolam group), 25 patients received midazolam. In group B (dexmedetomidine group), 25 patients received dexmedetomidine.

DETAILED DESCRIPTION:
Background: Peribulbar blocks are commonly used for cataract surgery, providing effective anesthesia with reduced recovery time. The addition of sedative agents, such as dexmedetomidine or midazolam, may enhance the anesthetic effect and patient comfort while maintaining hemodynamic stability. However, the optimal sedative agent for use in this context remains uncertain.

Objective: This study aimed to compare the efficacy and safety of dexmedetomidine and midazolam as adjuvants to local anesthetic in peribulbar blocks for cataract surgery.

Methods: A randomized, double-blind clinical trial included 50 patients aged 18-75 years with the American Society of Anesthesiologists physical status I-II who were scheduled for cataract surgery under peribulbar block. Participants were randomly allocated to two groups: Group A received midazolam (1 mg), and Group B received dexmedetomidine (50 µg), combined with a standard mixture of local anesthetics. The primary outcomes included the onset and duration of motor and sensory block and lid akinesia. Secondary outcomes assessed the quality of motor and sensory block, lid akinesia using the Ocular Anesthesia Scoring System, sedation levels using the Ramsay Sedation Score, the occurrence of local or systemic complications, and satisfaction levels reported by both patients and surgeons.

Keywords: dexmedetomidine; midazolam; peribulbar block; cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cataract Disease
* Scheduled for cataract surgery
* American Society of Anesthesiologists physical status I or II.

Exclusion Criteria:

* History of allergy to any of the study medications
* Had impaired mental status
* Had coagulation abnormalities
* Had severe cardiac disease
* Had chronic obstructive lung disease
* Had a history of sleep apnea
* Refused to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
onset of motor block | Intraoperative from the moment of local anesthesia injection until the moment of complete and full globe akinesia up to 1 hour
  The period of time that passed after the local anesthetic mixture was injected before the eye globe was completely immobile

SECONDARY OUTCOMES:
onset of sensory block | Intraoperative from the moment of local anesthesia injection until the moment of complete insensitivity and absent reflexes of the eye up to 1 hour
  the period of time following the local anesthetic mixture injection that resulted in total insensitivity and absent eye reflexes
length of the motor block | Periperative from the moment of complete and full globe akinesia until the moment of return back of eye movement up to 1 hour
  The time it takes for the entire eye globe to return to free motion after experiencing akinesia
length of the sensory block | Periperative from the moment of complete areflexia until the moment of return back of sensation and reflexes up to 1 hour
  The amount of time before the entire eye globe regains sensation after experiencing insensitivity and areflexia andreflexes

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrhman Alshawadfy, MD, Principal Investigator — Suez Canal University
Locations (1):
- Suez canal university, Ismailia, Egypt